CLINICAL TRIAL: NCT03201731
Title: Social Isolation and Loneliness in Very Late-onset Schizophrenia-like Psychosis: A Case-control Study
Brief Title: Social Isolation and Loneliness in Older People
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 17/0347
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Very Late Onset Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Those diagnosed with a non-organic, non-affective psychotic disorder for the first time after age 60, recruited from a Community Mental Health Team.
- Controls: Those aged 60 and above in contact with the same Community Mental Health Team for another mental health problem aside from a psychotic disorder or dementia.

SUMMARY:
Although psychotic disorders such as schizophrenia usually present in late adolescence or early adulthood, research suggests that a substantial subset of people are diagnosed for the first time after the age of 60. This condition is referred to as 'very late-onset schizophrenia-like psychosis' (VLOSLP). People with VLOSLP are thought to experience high levels of social isolation, yet there has been little research systematically examining this. Additionally, little is known about how lonely people with VLOSLP feel, or how this group relate to and perceive other people.

This study aims to examine levels of social isolation and loneliness in patients with VLOSLP. The investigators also aim to explore aspects of social cognition in relation to VLOSLP.

A case-control study design will be used to examine the relationship between VLOSLP, loneliness, social isolation and social cognition. The case group will be people diagnosed with a non-organic psychotic disorder after age 60. The comparison group will be those aged 60 and above in contact with mental health services for a mental health difficulty, except from a psychotic disorder or dementia.

ELIGIBILITY:
Cases

Inclusion criteria:

* Aged 60 and above.
* Diagnosed with a psychotic disorder after age 60.

Exclusion criteria:

* Diagnosed with a psychotic disorder before age 60.
* Dementia diagnosis.
* Mild cognitive impairment diagnosis.
* Clear organic cause for psychosis.
* Does not speak English to the degree needed to engage with study materials.
* Mental health problems too severe to fully engage with the study.
* Other medical or psychosocial factor that could limit ability to fully engage with study materials, such as severe intellectual disability or imminently life-limiting illness.

Controls

Inclusion criteria:

* Aged 60 and above.
* Diagnosed with any mental health disorder except from a psychotic disorder, dementia, or severe depression.

Exclusion criteria:

* Diagnosed psychotic disorder, drug-induced psychosis or organic psychosis.
* Dementia diagnosis.
* Mental health problems too severe to fully engage with the study.
* Does not speak English to the degree needed to engage with study materials.
* Other medical or psychosocial factor that could limit ability to fully engage with study materials, such as severe intellectual disability or imminently life-limiting illness.

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cases and controls will be recruited from the same Community Mental Health Team.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
UCLA loneliness Scale (version 3) (Russel, 1996) | Total assessment time: two hours
  The UCLA loneliness scale is a 20-item measure of subjective feelings of loneliness. The scale has been validated for use in the elderly. Each item is scored from 1 (never) to 4 (often). Items include 'I lack companionship' and 'People are around me but not with me'. The scale yields an overall loneliness score between 0-80.
Lubben Social Network Scale - 6 (LSNS-6) (Lubben et al., 2006) | Total assessment time: two hours
  The LSNS-6 is a six-item self-report scale to assess social isolation in older adults by measuring perceived social support received from family and friends. The scale assesses the size, closeness and frequency of contacts within a respondent's social network, with a subscale for friends and another for family. Higher scores indicate larger social networks and lower scores indicate higher levels of social isolation. Questions include 'How many relatives do you see or hear from at least once a month?' and 'How many friends do you feel at ease with that you can talk about private matters?'.

SECONDARY OUTCOMES:
Ambiguous Intentions Attribution Questionnaire (Combs, Penn, Wicher & Waldheter, 2007) | Total assessment time: two hours
  This questionnaire is designed to examine attribution bias with a particular focus on hostile social-cognitive bias. The researcher will read participants each vignette and ask them to imagine that the scenario is happening to them. Participants rate whether the action was performed on purpose, with ratings from 1 (definitely no) to 6 (definitely yes), how angry it would make them feel from 1 (not at all angry) to 5 (very angry) and how much they would blame the other person from 1 (not at all) to 5 (very much). These are totaled to create an overall score. Responses to each item are averaged across scenarios and summed, with higher scores indicating greater blame.
The Faux Pas test (Stone, Baron-Cohen & Knight, 1998) | Total assessment time: two hours
  The Faux Pas test is designed to measure theory of mind, or the ability to make inferences about the thoughts, beliefs and intentions of others and to understand the possible motivations underlying others' actions. In this test, theory of mind is measured using short vignettes followed by a series of questions. We shall use a short version of the test developed by Negrão et al., (2016). This test uses 5/10 faux pas stories and 5/10 control stories from the original Faux Pas Test. After each story is read, participants will be asked five questions for: detecting a faux pas, understanding the faux pas, understanding the mental state of the faux pas recipient, understanding the mental state of the person delivering the faux pas and understanding the details but without making inferences about the mental states of the characters in the story.